CLINICAL TRIAL: NCT04875455
Title: Development of a Database (Register) for Quality Assurance and Optimization of the Postoperative Results of Premium Intraocular Lenses
Brief Title: Premium Trifocal IOL Comparative Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY1705
Record Dates: First submitted 2021-05-01; First posted 2021-05-06 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Cataract; Lens Opacities; Presbyopia
Keywords: Intraocular lens; Trifocal
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Intervention Model Description: Study procedure guidelines
  Patients who were previously treated with a premium IOL (Panoptix, POD FGF, POD F) are continuously included:
  Retrospective:
  Routine data collected up to the first study visit (preoperative, intraoperative and postoperative) are evaluated retrospectively
  Prospective:
  2-4 months postoperatively: refraction and vision, slit lamp and fundus examination, intraocular
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: POD F GF (BVI Medical), POD F (BVI Medical), Panoptix (Alcon Inc) IOL implantation (Experimental): PhysIOL POD F GF: 50 (bilateral implantation) PhysIOL POD F: 50 (bilateral implantation) Alcon PanOptix: 20 (bilateral implantation) In this study, patients have already received treatment, after receiving the consent, the routinely collected pre-, intra- and postoperative data will be pseudonymized and evaluated.
  Interventions: Device: POD F GF (BVI Medical), POD F (BVI Medical), Panoptix (Alcon Inc) IOL implantation

INTERVENTIONS:
Device: POD F GF (BVI Medical), POD F (BVI Medical), Panoptix (Alcon Inc) IOL implantation — In this study, patients have already received treatment, after receiving the consent, the routinely collected pre-, intra- and postoperative data will be pseudonymized and evaluated.

SUMMARY:
Short and long-term analysis of the refraction correction and optical image quality of modern premium intraocular lenses (IOLs) with the establishment of a database for quality assurance and optimization the computation constants of the lens power.

DETAILED DESCRIPTION:
Since the investigational lens, like conventional IOLs, is a posterior chamber lens which is widely implanted following cataract extraction, phacoemulsification is adopted. To assess the binocular vision, the investigational lens will be mono- or bilaterally implanted.

Clinically retro- and prospective, non-randomized, uncontrolled, open study at several centers: University Eye Clinic Heidelberg (leading center), Practice Center Ahaus in the Eye Clinic Ahaus, Breyer, Kaymak & Klabe Eye Surgery in Düsseldorf, nordBLICK Eye Center Kiel.

Main objectives:

1. Functional results (refraction and visual acuity results) Secondary goals:
2. Deviation target vs. achieved postoperative refraction (for constant optimization of the IOL calculation)
3. Subjective patient satisfaction
4. Visual quality (e.g. scattered light, contrast vision, spherical aberrations)
5. Stability of the results achieved postoperatively

ELIGIBILITY:
Inclusion criteria

* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Bilateral implantation of one of the following IOL models
* Alcon PanOptix (TFNT00)
* PhysIOL FineVision (POD F)
* PhysIOL FineVision (POD F GF)
* Uneventful cataract surgery with first clinical outcomes in the expected range
* Patient included in Premium IOL study protocol by signed informed consent

Exclusion criteria

* Age of patient <45 years
* Irregular astigmatism
* Postoperative manifested astigmatism of >1.0 D
* Difficulty for cooperation (distance from their home, general health condition)
* Clinically significant glaucoma
* Clinically significant macular degeneration, clinically significant macular edema or proliferative diabetic retinopathy
* Patients with keratoconus or keratectasia
* Any ocular comorbidity having a significant effect on the postoperative clinical outcomes
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalitis (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* AMD
* Intraoperative complications like capsular rupture etc.
* Patients who do not give informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Monocular Best corrected distance visual acuity (5 m) | Postoperative Day 75-105 (3 months)
  CDVA measured with ETDRS charts placed in 5m distance with best aided corrective glasses according to ISO 11979-7:2014.

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Auffarth, MD, PhD, Principal Investigator — University Hospital Heidelberg
Locations (4):
- Germany (4):
  - Augenklinik Ahaus, Ahaus
  - Internationale Innovative Ophthalmochirgie, Düsseldorf
  - Universitäts-Augenklinik Heidelberg, Heidelberg
  - Augentagesklinik Rheine, Rheine

IPD SHARING:
Plan to Share IPD: No